CLINICAL TRIAL: NCT06597201
Title: Multicenter, Prospective, Open-label, Randomized, Parallel-group Clinical Trial to Evaluate the Efficacy and Safety of Amino Acid (15) Peritoneal Dialysis Solution in Peritoneal Dialysis Patients with Malnutrition.
Brief Title: Evaluate the Efficacy and Safety of Amino Acid (15) Peritoneal Dialysis Solution in Peritoneal Dialysis Patients with Malnutrition.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chengdu Qingshan Likang Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAD-QSLK-401
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: End stage renal disease; peritoneal dialysis solution; malnutrition
MeSH Terms: conditions — Kidney Failure, Chronic; Malnutrition | interventions — Amino Acids; Dialysis Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Subjects were treated with 1 bag of amino acid (15) peritoneal dialysate (2L) once every morning, and then with conventional glucose peritoneal dialysate (lactate).
  Interventions: Drug: amino acid (15) peritoneal dialysis solution
- control group (Active Comparator): Subjects received conventional treatment with glucose peritoneal dialysis solution (lactate), which must include 1.5% glucose peritoneal dialysate (lactate) (2L) once.
  Interventions: Drug: glucose peritoneal dialysis solution

INTERVENTIONS:
Drug: amino acid (15) peritoneal dialysis solution — Subjects were treated with 1 bag of amino acid (15) peritoneal dialysis solution (2L) once every morning, and then with conventional glucose peritoneal dialysate (lactate).
  Arms: experimental group
Drug: glucose peritoneal dialysis solution — Subjects received conventional treatment with glucose peritoneal dialysis solution (lactate), which must include 1.5% glucose peritoneal dialysate (lactate) (2L) once.
  Arms: control group

SUMMARY:
This is a multicenter, randomized, parallel controlled Phase IV clinical study to evaluate the safety and efficacy of amino acid (15) peritoneal dialysis solution in patients undergoing peritoneal dialysis with malnutrition in CAPD patients undergoing peritoneal dialysis maintenance.

DETAILED DESCRIPTION:
After the subjects signed the informed consent, they entered the screening period (D-28 to D-1) for corresponding examination. Participants who were successfully screened were examined at baseline (D-3 to D-1) to re-verify the inclusion criteria. After re-verification of successful screening subjects, they were enrolled in 1:1 parallel groups according to the research center: experimental group treated with amino acid (15) peritoneal dialysate; Control group - glucose peritoneal dialysate treatment. Subjects were randomly enrolled and given the experimental drug from the next morning according to the randomized results. Subjects in the experimental group were treated with 1 bag of amino acid (15) peritoneal dialysate (2L) once a day in the morning, and were subsequently treated with conventional glucose peritoneal dialysate (lactate). Control subjects received conventional treatment with glucose peritoneal dialysis solution (lactate), which must include 1.5% glucose peritoneal dialysis solution (lactate) (2L) once. The number of peritoneal dialysate exchange, the amount of fluid exchange and the duration of abdominal retention were adjusted by the researchers according to the specific conditions of the patients. Efficacy and safety were observed during the treatment period (D1-D90). Blood routine and blood biochemistry were monitored for 30 days, 60 days and 90 days of treatment. nPNA, AMC, MAMC, SGA, BMI, Kt/V, etc. are monitored only at 90 days. The total daily ultrafiltration volume of the patients (the experimental group also recorded the ultrafiltration volume of amino acid peritoneal fluid), and all adverse events (aes) and serious adverse events (SAEs) were recorded in detail.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years of age (including 18 and 75 years of age), regardless of sex;
2. Stable CAPD patients treated with peritoneal dialysis for greater than or equal to 3 months;
3. 25 ≤ serum ALB ≤ 40 g/L on two consecutive occasions prior to enrollment (two occasions one week apart);
4. Blood potassium ≥ 3.5 mmol/L
5. C-reactive protein (CRP) ≤ 2 x upper limit of normal (ULN);
6. Carbon dioxide binding capacity >18 mmol/L;
7. Subjects voluntarily sign an informed consent form in writing prior to the commencement of any procedures related to the study, fully understand the purpose and significance of the trial, and are willing to comply with the trial protocol.

Exclusion Criteria:

1. Within the past 3 months prior to the screening period, there has been a history of peritonitis, other infections, or inflammatory diseases, with hospitalization records;
2. The possibility of receiving a kidney transplant during the study period;
3. Patients with inadequate dialysis and screening period kt/v<1.4;
4. Patients with hemoglobin less than 80g/L during the screening period;
5. Patients who have used amino acid (15) peritoneal dialysate within 6 months prior to the screening period.
6. Patients with bleeding events (active gastrointestinal hemorrhage, cerebral hemorrhage), cardiovascular and cerebrovascular events (cerebral infarction, myocardial infarction, etc., and NYHA grade ≥3 of cardiac function) within 30 days before screening period.
7. In patients with active diarrhea during the screening period, as assessed by investigators, affecting nutrient absorption(Except for patients with chronic diarrhea, stool frequency < 3 times/day);
8. patients with contraindications to amino acid (15) peritoneal dialysis solutions: 1) hypersensitivity to any of the components of the product; 2) Serum urea level >38 mmol/l; 3) Presence of uremic symptoms such as marked loss of appetite, nausea and vomiting at the time of screening; 4) Various inborn abnormalities of amino acid metabolism; 5) hepatic insufficiency (active hepatitis); active hepatitis B or C, cirrhosis, active liver disease or positive seropositivity for human immunodeficiency virus (HIV) within 6 months prior to screening; 6) Uncorrectable mechanical defects that the investigator assesses as affecting efficacy or increasing the risk of infection; 7) History of loss of peritoneal function or impairment of peritoneal function due to extensive adhesions;
9. Suffers from a malignant tumor or has a life expectancy of <6 months;
10. Routine daily use of 4.25% glucose dialysis solution during the screening period;
11. Diabetic subjects with poor prior glycemic control, e.g., HbAlc > 8%;
12. Women during pregnancy or breastfeeding;
13. Other circumstances that, in the opinion of the investigator, may make participation in this study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-06-29 (Estimated); Study Completion 2025-06-29 (Estimated)

PRIMARY OUTCOMES:
ALB | After 90 days of treatment
  To compare the difference in change from baseline in serum albumin (ALB) after 90 days of treatment of CAPD patients with amino acid (15) peritoneal dialysis solution versus conventional glucose peritoneal dialysis solution (lactate).

SECONDARY OUTCOMES:
serum transferrin | After 30, 60, and 90 days of treatment
  To compare the changes of serum transferrin in CAPD patients treated with amino acid (15) peritoneal dialysate and conventional glucose peritoneal dialysate (lactate) at 30 days, 60 days and 90 days compared with baseline.
arm muscle circumference (AMC) | After 90 days of treatment
  omparison of standardized upper arm muscle circumference (AMC) changes from baseline after fasting peritoneal dialysis fluid emptying between amino acid (15) peritoneal dialysis solution and conventional glucose peritoneal dialysis solution (lactate) in CAPD patients treated for 90 days.
standardized protein nitrogen occurrence rate (nPNA) | After 90 days of treatment
  To compare the change of standardized protein nitrogen occurrence rate (nPNA) in CAPD patients treated with amino acid (15) peritoneal dialysis solution and conventional glucose peritoneal dialysis solution (lactate) after 90 days from baseline.
subjective comprehensive nutritional assessment (SGA) | After 90 days of treatment
  To compare the change of subjective comprehensive nutritional assessment (SGA) in CAPD patients treated with amino acid (15) peritoneal dialysis solution and conventional glucose peritoneal dialysis solution (lactate) after 90 days from baseline.
middle arm muscle circumference (MAMC) | After 90 days of treatment
  To compare the change of middle arm muscle circumference (MAMC) in CAPD patients treated with amino acid (15) peritoneal dialysis solution and conventional glucose peritoneal dialysis solution (lactate) after 90 days from baseline.
serum prealbumin | After 30, 60, and 90 days of treatment
  To compare the changes of serum prealbumin in CAPD patients treated with amino acid (15) peritoneal dialysate and conventional glucose peritoneal dialysate (lactate) at 30 days, 60 days and 90 days compared with baseline.
serum albumin | After 30, 60, and 90 days of treatment
  To compare the changes of serum albumin in CAPD patients treated with amino acid (15) peritoneal dialysate and conventional glucose peritoneal dialysate (lactate) at 30 days, 60 days and 90 days compared with baseline.
body mass index (BMI) | After 90 days of treatment
  To compare the change of standardized protein nitrogen occurrence rate (nPNA) in CAPD patients treated with amino acid (15) peritoneal dialysis solution and conventional glucose peritoneal dialysis solution (lactate) after 90 days from baseline.

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University People&'s Hospital, Beijing, Beijing Municipality
  - Wuhan NO.1 Hospital, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Ganzhou People's Hospital, Ganzhou
  - Affiliated Hospital of Guangdong Medical University, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The Affiliated Hospital of Southwest Medical University, Luzhou
  - Meishan Hospital, West China Hospital, Sichuan University (Meishan People's Hospital), Meishan
  - Jiangsu Province Hosipital, Nanjing
  - The Affiliated Hospital of Nanjing university Medical School, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Shanghai Sixth People's Hospital Affiliated to Shanghai JiaoTong University, Shanghai
  - General Hospital of Northern Theater Command, Shenyang
  - The Central Hospital of Wuhan, Wuhan
  - Zhongshan Hospital Xiamen University, Xiamen
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang
  - The Second People's Hospital of Yibin City, Yibin
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] My Thuc LT, Dung NQ, Ha VN, Tam ND, Hang Nga NT. Actual diet and nutritional deficiencies status in children on peritoneal dialysis at the Vietnam National Hospital of Pediatrics. Saudi J Kidney Dis Transpl. 2019 Jul-Aug;30(4):924-931. doi: 10.4103/1319-2442.265470. PMID 31464251
- [Background] Kopple JD, Bernard D, Messana J, Swartz R, Bergstrom J, Lindholm B, Lim V, Brunori G, Leiserowitz M, Bier DM, et al. Treatment of malnourished CAPD patients with an amino acid based dialysate. Kidney Int. 1995 Apr;47(4):1148-57. doi: 10.1038/ki.1995.164. PMID 7783413
- [Background] Tjiong HL, Swart R, van den Berg JW, Fieren MW. Amino Acid-based peritoneal dialysis solutions for malnutrition: new perspectives. Perit Dial Int. 2009 Jul-Aug;29(4):384-93. PMID 19602603